CLINICAL TRIAL: NCT01644383
Title: Meaning in Life of Youth Infected With HIV
Brief Title: Meaning of Life in HIV-infected Youths
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Chulalongkorn University (Other); Pediatric department, Chulalongkorn University, Bangkok, Thailand (Unknown); SEARCH Research Foundation (Other); Wayne State University (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: HIV-NAT 109
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Meaning of Life
Keywords: meaning of life; logotherapy; HIV-infected teenagers; adherence
MeSH Terms: interventions — Logotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment arm (logotherapy) (Experimental): Participants in Arm I will attend the logotherapy group sessions by the trained psychologist for 4 visits (see Table II, III). The number of participants in group sessions will be 20 participants per group.
  Interventions: Behavioral: logotherapy
- Control arm (general health education) (No Intervention): Participants in Arm II will attend the routine health education by the nurse. The number of participants in group session will be 20 participants per group.

INTERVENTIONS:
Behavioral: logotherapy — Logotherapy is therapy during which the interaction between the therapist and the client centres on the topic of meaning. The problems that the clients experience are presented to the client as inseparable parts of his everyday life. The client is then challenged to discover his/her meaning and to take responsibility in facing up to his/her problem. This approach is aimed at helping the client to deal and understand what his /her existences entail.
  Arms: Treatment arm (logotherapy)

SUMMARY:
Logotherapy has never been evaluated in HIV-infected teenagers. In this study, we will evaluate the meaning of life by using The Purpose in Life Test and the affect of logotherapy in HIV infected youth at HIV-NAT, Thai Red Cross AIDS Research Centre and King Chulalongkorn Memorial Hospital.

DETAILED DESCRIPTION:
In the HAART era, HIV infected children can live longer and will grow up to become teenagers. However, some may develop psychosocial problems because they have lost family members, experienced poverty, social discrimination etc. Being a normal teenager is tough and is the most complex period of his/her life. This is the period when most teenagers will find their identity and reasons for living. Therefore it is believed that interventions may help HIV-infected teenagers better deal with life. For this study, logotherapy, a therapy that will help a person to discover his/her purpose in life, live meaningful life, and attain self-esteem was used. The success of the intervention was evaluated by using The Purpose in Life Test.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16-24 years
2. HIV seropositive
3. HIV disclosed
4. Understand Thai language
5. Parent signed written informed consent

Exclusion Criteria:

1. Mental or psychological disorder or having active suicidal idea or attempt
2. Having no permanent address

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2011-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
PIL score | week 48
  Change of PIL score at baseline and follow up visit between the two arms

SECONDARY OUTCOMES:
QOL | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arunya Tuicomepee, PhD, Principal Investigator — Chulalongkorn University
Locations (1):
- HIV-NAT, the Thai Red Cross AIDS Research Centre, Bangkok, Thailand

REFERENCES:
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org